CLINICAL TRIAL: NCT03807843
Title: Phase 2 Study of a Live Attenuated Measles Virus-Vectored Chikungunya Vaccine in Previously Exposed Adults
Brief Title: Chikungunya Vaccine (V184) Study in Previously Exposed Adults (V184-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V184-006; MV-CHIK-206 (Other: Themisbio)
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, randomized, double-blinded, interventional, safety study
Who Masked: Participant, Investigator
Masking Description: Study medication is available as liquid frozen vaccine product or saline for injection (placebo). The actual study injections will be forwarded to the investigator (injector) in a blinded fashion (injection ready syringes containing either vaccine or placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V184 (Experimental): Participants will receive 2 vaccinations with V184 administered via intramuscular (IM) injection at 5 × 10^5 Tissue Culture Infectious Dose (TCID50) per dose on Days 0 and 28.
  Interventions: Biological: V184
- Placebo (Placebo Comparator): Participants will receive 2 injections of sterile physiological saline administered via IM injection on Days 0 and 28.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: V184 — Recombinant live Schwarz-strain measles-vectored vaccine expressing chikungunya virus structural proteins. Liquid frozen, life attenuated, measles vectored V184 vaccine administered via IM injection at 5 × 10^5 TCID50 (+/- 0.5 log) per dose.
  Other Names: MV-CHIK; MV-CHIK vaccine; MV-CHIK/DP (drug product)
  Arms: V184
Other: Placebo — Sterile physiological saline for IM injection
  Arms: Placebo

SUMMARY:
Safety and immunogenicity of the investigational V184 chikungunya vaccine will be tested in participants with history of chikungunya infection. Initially 21 to 50 year old participants will be enrolled; after favorable review of safety data, participants aged 51 to 65 will be enrolled.

DETAILED DESCRIPTION:
This will be a randomized double-blind interventional clinical study. This study proposes to evaluate the safety and immunogenicity of the investigational V184 live recombinant measles-vectored chikungunya vaccine delivered in 2 vaccinations, 28 days apart compared with saline placebo. After providing informed consent, individuals will be screened for eligibility including verification of previous exposure to chikungunya virus. They will then be randomized in a double-blind fashion to receive either V184 or saline placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Previous infection with chikungunya as verified by a serum immunoassay.
* Able to provide informed consent.
* Available and accessible for the duration of the trial.
* Able and willing to comply with all requirements of the study.
* For women of childbearing potential, willing to practice adequate contraception for the duration of the study.
* Medical history and physical examination findings are considered normal or not clinically significant in the opinion of the Investigator, which includes resolution of any arthralgias that may have occurred during prior chikungunya infection, as well as the absence of synovitis.
* Laboratory values are considered normal or not clinically significant in the opinion of the Investigator. If laboratory screening tests are out of the normal reference range and of potential clinical significance, the test(s) may be repeated up to 2 times (a total of 3 per screening evaluation) at the discretion of the Investigator, and the repeat values and their potential clinical significance will be used to determine eligibility.
* History of immunity to measles. For persons born after 1957, this will be established by a history of compliance with vaccination policies that included measles vaccination or known vaccination as an adult at least one month before they are randomized. Volunteers born before 1957 will be presumed to have immunity to measles based on natural exposure in accordance with US Centers for Disease Control and Prevention (CDC) guidelines [McLean 2013].

Exclusion Criteria:

* Taking medication or other treatment for unresolved symptoms attributed to a previous chikungunya virus infection.
* Prior receipt of any investigational chikungunya or other alphavirus vaccine. To date, no alphavirus vaccines have been commercially available in the United States.
* Recent infection:

  * self-limited upper respiratory infections until afebrile without medication for >1 week;
  * chikungunya unless/until asymptomatic (other than mild subjective symptoms not requiring treatment) for >3 months;
  * non-recurrent upper respiratory or urinary tract infections successfully treated with antibiotics, until asymptomatic for 1 month after full antibiotic course has been completed.
* History of an acute allergic or anaphylactic reaction to any vaccine.
* History of an immunosuppressive disorder (such as human immunodeficiency virus [HIV] infection, Common Variable Immune Deficiency), chronic infection (such as chronic hepatitis B or C), autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune thyroid disease), or any medical condition that, in the opinion of the Investigator, could lead to an atypical immune response to the vaccine.
* History of moderate or severe non-traumatic arthritis or arthralgia within 3 months of the Screening Visit.
* Recent (within 30 days), current or anticipated use of any immunosuppressive or immune modifying medication including corticosteroids (excluding nasal, ophthalmic, and other topical preparations).
* Other vaccination or planned vaccination within 4 weeks of either study dose (seasonal influenza vaccine excepted).
* Receipt or planned receipt of blood products including immunoglobulins within 120 days of the Screening Visit.
* Pregnant or lactating or planning pregnancy during the trial.
* Known alcohol or other substance abuse that in the opinion of the Investigator affects the ability or willingness of the participant to understand and comply with the study protocol.
* Participation in another clinical study within the past 30 days in which the participant was exposed to an investigational product (pharmaceutical product or placebo or device) or planned participation in another interventional clinical study while participating in this study.
* Relevant history of any medical condition that, in the opinion of the Investigator, may interfere with the safety of the participant or aims of the study.
* History of neoplastic disease (excluding successfully treated non-melanoma skin cancer or cervical intraepithelial neoplasia) within the past 5 years or a history of any hematological malignancy.
* Behavioral or psychiatric disease or cognitive impairment that in the opinion of the Investigator affects the ability or willingness of the participant to understand and comply with the study protocol.
* Non-consent to storage of blood specimens for future research.
* Persons in direct relationship with the Sponsor or its contracted service providers, the contract research organisation (CRO) or its subcontractors, the Investigator, or study site staff. Direct relationship includes first degree relatives or dependents (children, spouse/partner, siblings or parents), as well as employees (site or Sponsor).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- San Juan Hospital, Research Unit, San Juan, Puert Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- V184: Participants received 2 vaccinations with V184 administered via intramuscular (IM) injection at 5 × 10^5 Tissue Culture Infectious Dose (TCID50) per dose on Days 0 and 28.
- Placebo: Participants received 2 injections of sterile physiological saline administered via IM injection on Days 0 and 28.
Period: Overall Study
Arm/Group | V184 | Placebo
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V184 | Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.29) | 37.3 (11.37) | 39.3 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 41
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence temporally associated with the use of the treatment that did not necessarily have a causal relationship with the treatment. "Solicited AEs" included fever, fatigue, headache, malaise, myalgia, nausea/vomiting, joint pain or injection site itching, pain/tenderness, erythema/redness or induration/swelling that occurred within 7 days of vaccination. The number of participants with solicited AEs following Vaccination 1 (Day 0) or Vaccination 2 (Day 28) were reported for each group.
Time Frame: Up to 7 days after vaccination (up to Day 35)
Population: All participants that received at least one dose of vaccine/placebo were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | V184 | Placebo
Number analyzed (Participants) | 21 | 20
Participants | 15 | 11

2. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Serum Neutralizing Antibodies (nAb) to V184 Over Time
Description: Serum samples were collected and the titers of serum neutralization antibodies were assessed. GMTs were calculated using a mixed effects model with treatment (V184 versus placebo), visit and age group, and treatment visit interaction as fixed factors and participant as a random effect. GMFR was defined as the geometric mean of the ratio of concentration at specified timepoints after vaccination divided by concentration at baseline (Day 0).
Time Frame: Days 0, 28, 56, and 196
Population: All participants that received both doses of vaccine/placebo, had at least one post-vaccination immunogenicity assessment, and did not experience a protocol deviation that affected their immunogenicity evaluation were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V184 | Placebo
Number analyzed (Participants) | 18 | 17
Ratio
  Day 28 | 1.5 [1.2 to 1.8] | 0.9 [0.7 to 1.2]
  Day 56: number analyzed (Participants) | 17 | 17
  Day 56 | 1.9 [1.5 to 2.3] | 0.9 [0.7 to 1.1]
  Day 196: number analyzed (Participants) | 17 | 17
  Day 196 | 1.3 [1.0 to 1.6] | 1.0 [0.8 to 1.3]
Statistical Analysis 1: Comparison: V184 vs Placebo; Day 28 V184 GMFR/Placebo GMFR Ratio The ratio of V184 GMFR/Placebo GMFR at Day 28 was derived from the mixed effects model used to determine GMFR; Test type: Other; p = 0.004, Mixed Effects Model; V184 GMFR/Placebo GMFR Ratio = 1.6, 95% CI 2-sided [1.2 to 2.1]
Statistical Analysis 2: Comparison: V184 vs Placebo; Day 56 V184 GMFR/Placebo GMFR Ratio The ratio of V184 GMFR/Placebo GMFR at Day 56 was derived from the mixed effects model used to determine GMFR; Test type: Other; p < 0.001, Mixed Effects Model; V184 GMFR/Placebo GMFR Ratio = 2.1, 95% CI 2-sided [1.5 to 2.8]
Statistical Analysis 3: Comparison: V184 vs Placebo; Day 196 V184 GMFR/Placebo GMFR Ratio The ratio of V184 GMFR/Placebo GMFR at Day 196 was derived from the mixed effects model used to determine GMFR; Test type: Other; p = 0.121, Mixed Effects Model; V184 GMFR/Placebo GMFR Ratio = 1.3, 95% CI 2-sided [0.9 to 1.7]

3. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence temporally associated with the use of the treatment that did not necessarily have a causal relationship with the treatment. "Unsolicited AEs" were defined as events reported within 7 days after each vaccination and not defined as solicited AE, and all AEs reported more than 7 days after vaccination. The number of participants with unsolicited AEs were reported for each group.
Time Frame: Up to Day 196
Population: All participants that received at least one dose of vaccine/placebo were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | V184 | Placebo
Number analyzed (Participants) | 21 | 20
Participants | 3 | 3

4. Primary Outcome: Number of Participants With Solicited and Unsolicited AEs of Grade 2 or Higher According to the 2007 Toxicity Grading Scale for Healthy Adult Volunteers Enrolled in Preventive Vaccine Clinical Trials (2007)
Description: An AE was defined as any untoward medical occurrence temporally associated with the use of the treatment that did not necessarily have a causal relationship with the treatment. "Solicited AEs" included fever, fatigue, headache, malaise, myalgia, nausea/vomiting, joint pain or injection site itching, pain/tenderness, erythema/redness or induration/swelling that occurred within 7 days of vaccination. "Unsolicited AEs" were defined as events reported within 7 days after each vaccination and not defined as solicited AE, and all AEs reported more than 7 days after vaccination. AEs were graded by the investigator for severity as per the FDA Toxicity Grading Scale for Healthy Adults Enrolled in Vaccine Clinical Trials (2007), where Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=potentially life threatening. A higher grade indicates increased severity of AE. The number of participants with solicited and unsolicited AEs of grade 2 (moderate) or higher were reported for each group.
Time Frame: Up to Day 196
Population: All participants that received at least one dose of vaccine/placebo were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | V184 | Placebo
Number analyzed (Participants) | 21 | 20
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to Day 196
Description: All-Cause Mortality table includes all randomized participants. Serious and Other AE tables include all randomized participants who received at least 1 dose of study treatment.
Arm/Group | V184 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 17/21 | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V184 (N=21) | Placebo (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (4) | 6 (9)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 11 (17) | 5 (10)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 5 (8)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the Investigator may prepare a joint publication with the Sponsor and Project Oversight Agency. The Investigator must not submit any part of the data from this protocol for publication without the prior consent of the Sponsor and Project Oversight Agency.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03807843/Prot_SAP_000.pdf